CLINICAL TRIAL: NCT05787015
Title: Testing a Personalized Normative Feedback Intervention for Vaccine Hesitancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Scott Graupensperger, Assistant Professor, Department of Psychiatry and Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00015728; 6NU87PS004366-03-02 (Other Grant/Funding Number: Center for Disease Control and Prevention)
Record Dates: First submitted 2023-03-03; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: COVID-19; Vaccine Hesitancy
MeSH Terms: conditions — COVID-19; Vaccination Hesitancy | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine Norms Feedback (Experimental): The participants in the treatment condition will receive personalized normative feedback (PNF) that entails correcting normative misperceptions for US young adults' vaccine uptake rates and prevalence of vaccine hesitancies (e.g., fear of side effects). Participants will be shown discrepancies between their perceived estimate of young adults' vaccination rates and actual national estimates derived from the US Census Bureau's Household Pulse Survey to highlight, in most cases, that they underestimated the vaccination norms.
  Interventions: Behavioral: Vaccine Norms Feedback
- Alcohol Norms Feedback (Active Comparator): Participants randomized to control will complete all measures at the same time as participants in the treatment condition, but will not receive any normative information regarding vaccines. Instead, to match for attention and provide potential benefit, those in the control condition will receive a standard dynamic norms feedback pertaining to alcohol use norms and behaviors.
  Interventions: Behavioral: Alcohol Norms Feedback

INTERVENTIONS:
Behavioral: Vaccine Norms Feedback — Personalized normative feedback pertaining to normative misperceptions about vaccination rates and hesitant attitudes.
  Arms: Vaccine Norms Feedback
Behavioral: Alcohol Norms Feedback — Personalized normative feedback pertaining to normative misperceptions about alcohol use.
  Arms: Alcohol Norms Feedback

SUMMARY:
Rationale: The highest rates of coronavirus disease (i.e., COVID-19) vaccine hesitancy in the US are among young adults (YAs) aged 18-25. Our preliminary studies show that social norms - perceptions of peers' vaccination attitudes/behaviors - are most strongly related to YAs' vaccine intentions/uptake. Most YAs underestimate the perceived importance of vaccination and their peers' intentions to be vaccinated. The proposed research will develop and test an intervention to correct misperceived norms for vaccination hesitancy and uptake.

Methodology: Rapid prototyping with 20 unvaccinated YAs will help refine the content and design of the online intervention. Then, a diverse national sample (N=600) of unvaccinated YAs will be randomized to treatment or an attention-matched control. The treatment condition will receive personalized normative feedback (PNF) designed to correct normative misperceptions for vaccine hesitancy and uptake.

Normative feedback will be derived from the US Census Bureau's Household Pulse Survey. Follow-up surveys will be administered at 1, 2, 3, and 6 months to assess key outcomes including vaccine uptake, intentions, and reasons for vaccine hesitancy.

Aims and Data Analysis:

* Aim 1: Develop and refine a PNF intervention for vaccine hesitancy/uptake with user feedback from YAs. Rapid analysis of qualitative data will involve looking for themes in responses. Changes will be made iteratively to refine intervention content, design, and delivery.
* Aim 2: Evaluate intervention efficacy for increasing vaccine uptake and reducing time to first vaccine dose, relative to control, over the following year.
* Aim 3: Examine mediators (changes in perceived norms) and moderators (intellectual humility, identification with other people and young adults) of intervention efficacy. A longitudinal moderated mediation model will be examined.

Impact: Findings will clarify the causal role of psychological determinants of vaccine hesitancy (social norms, intellectual humility, group identification). If preliminary intervention efficacy is supported, this intervention could be a low-cost, and easily disseminated strategy to promote YAs' vaccine uptake and contribute to public health efforts to address the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* 18-24 years old (at screening)
* Reside in the United States.
* Have not received a COVID-19 vaccine (at screening)
* Pass attention checks.

Exclusion Criteria:

* Not meeting inclusion criteria.
* Not fluent in English.
* Not providing consent.
* Unwilling to participate.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
COVID-19 vaccine uptake | Through study completion, an average of 6 months
  Proportion of participants that have received a COVID-19 vaccine, following intervention
COVID-19 vaccine attitudes | Through study completion, an average of 6 months
  Attitudes towards receiving a COVID-19 vaccine measured using the Vaccination Attitudes Examination Scale (modified to COVID-19 vaccines).

CONTACTS AND LOCATIONS:
Overall Officials: Scott Graupensperger, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States